CLINICAL TRIAL: NCT03564678
Title: Mitochondrial Cofactors for the Treatment of Hyperbilirubinemia Due to PEG-Asparaginase and or Inotuzumab Ozogamicin in Patients With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Levocarnitine and Vitamin B Complex in Treating PEG-Asparaginase or Inotuzumab Ozogamicin-Induced Hyperbilirubinemia in Patients With Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request. Slow accrual and lack of clinical interest
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0978; NCI-2018-01253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0978 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-05-18; First posted 2018-06-21 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Hyperbilirubinemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hyperbilirubinemia | interventions — Carnitine; Vitamin B Complex; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (levocarnitine, vitamin B complex) (Experimental): Patients receive levocarnitine IV over 2-3 minutes every 6 hours up to 4 times a day (inpatient) or PO TID (outpatient). Patients also receive vitamin B complex PO BID. Treatment continues for up to 30 days after the last dose of either PEG-asparaginase or inotuzumab, or until Tbili of ≤ 1.5 x ULN or at least a 50% reduction in peak Tbili is achieved.
  Interventions: Dietary Supplement: Levocarnitine; Drug: Vitamin B Complex

INTERVENTIONS:
Dietary Supplement: Levocarnitine — Given IV
  Other Names: Carnitor; L-carnitine
Drug: Vitamin B Complex — Given PO
  Other Names: Becotin; Neurobion

SUMMARY:
This phase II trial studies how well levocarnitine and vitamin B complex works in treating abnormal high liver enzyme levels (hyperbilirubinemia) caused by treatment with PEG-asparaginase or inotuzumab ozogamicin in patients with acute lymphoblastic leukemia. Amino acids, such as levocarnitine, may work in normalizing liver enzyme levels due to treatment. Vitamin B complex is a dietary supplement that may be used for patients with nutritional deficiencies. Giving levocarnitine and vitamin B complex may work better in treating hyperbilirubinemia in patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Patients receive levocarnitine intravenously (IV) over 2-3 minutes every 6 hours up to 4 times a day (inpatient) or orally (PO) three times a day (TID) (outpatient). Patients also receive vitamin B complex PO twice daily (BID). Treatment continues for up to 30 days after the last dose of either PEG-asparaginase or inotuzumab, or until Tbili of ≤ 1.5 x ULN or at least a 50% reduction in peak Tbili is achieved.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Non-English speakers may be enrolled.
* Patients with a diagnosis of ALL who are receiving treatment with PEG-asparaginase or inotuzumab ozogamicin with Tbili > 3 x ULN
* Signed informed consent

Exclusion Criteria:

* Pregnant or nursing women
* Known hypersensitivity to levocarnitine or vitamin B complex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Levocarnitine, Vitamin B Complex)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Levocarnitine, Vitamin B Complex)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 41 [26 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Normalization of hyperbilirubinemia (Total bilirubin < 1.5 x ULN) or at least 50% reduction in peak total bilirubin within 11 days.
Time Frame: Up to 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Levocarnitine, Vitamin B Complex)
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Up to 6 years, 4 months and 28 days
Arm/Group | Treatment (Levocarnitine, Vitamin B Complex)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Levocarnitine, Vitamin B Complex) (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotranserase increased (Investigations) | 4 (5)
alkaline phos increased (Investigations) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Bacteremia (Infections and infestations) | 2 (2)
blood bilirubin increased (Investigations) | 5 (5)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
creatinine increased (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
herpes simplex reactivation (Infections and infestations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
ileal obstruction (Gastrointestinal disorders) | 1 (1)
INR increased (Investigations) | 5 (6)
lung infection (Infections and infestations) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
neutrophil count decreased (Investigations) | 8 (9)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 9 (10)
Serum amylase increased (Investigations) | 1 (1)
Lipase Increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03564678/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03564678/ICF_000.pdf